CLINICAL TRIAL: NCT01804283
Title: Effects of Ischemic Postconditioning on Expression of Apoptosis-related MicroRNAs and Genes in Human Double Valve Replacement
Brief Title: Effects of Ischemic Postconditioning on MicroRNAs in Double Valve Replacement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Central South University (Other)
Responsible Party: Principal Investigator, Luo Wanjun, Prof., Central South University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: CmiR-001
Record Dates: First submitted 2013-02-23; First posted 2013-03-05 (Estimated); Last update posted 2013-03-05 (Estimated); Status verified 2013-03

CONDITIONS: Cardiopulmonary Bypass; Ischemic Postconditioning
MeSH Terms: interventions — Ischemic Postconditioning; Heart-Lung Machine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CON (Sham Comparator): Patients undergoing double valve replacement (aortic and mitral).
  Interventions: Procedure: double valve replacement; Device: heart-lung machine; Device: Aortic cross-clamp
- IPO (Experimental): Patients undergoing double valve replacement (aortic and mitral) with ischemic postconditioning.
  Interventions: Procedure: ischemic postconditioning; Procedure: double valve replacement; Device: heart-lung machine; Device: Aortic cross-clamp

INTERVENTIONS:
Procedure: ischemic postconditioning — multiple brief ischemic-reperfusion episodes immediately after sustained ischemic insult
  Postconditioning was started at 30 s after aortic cross declamping, and the aorta was re-clamped for 30 s rendering global myocardial ischemia. Meanwhile aortic root suction was established during aortic re-clamping, and thereafter, the aortic clamp was released for 30 s for full myocardial reperfusion. The cycle was repeated three times after cardioplegic arrest.
  Arms: IPO
Procedure: double valve replacement — The double valve replacement is a procedure in which surgery is used to replace diseased aortic and mitral heart valves.
Device: heart-lung machine — The heart-lung machine is commonly used in open heart surgery including double valve replacement to support the circulation during the operation.
Device: Aortic cross-clamp — a surgical instrument used in cardiac surgery to clamp the aorta

SUMMARY:
1. Cardiopulmonary bypass and cardioplegic arrest could regulate expression of microRNAs in patients undergoing double valve replacement (aortic and mitral).
2. The modulation of myocardial microRNAs by cardiopulmonary bypass and cardioplegic arrest may be rescued by ischemic postconditioning.
3. Downstream effectors would also be affected.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive eight patients with rheumatic heart valve disease undergoing elective double valve replacement(aortic and mitral)are considered for participation in this study.

Exclusion Criteria:

* insulin-dependent diabetes mellitus
* pulmonary, renal, or hepatic failure
* infective valve disease
* valve disease with coronary artery disease
* hypertension
* emergency and reoperations
* received aspirin,corticosteroids, or statin preoperatively
* received preoperative inotropic support

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2013-03; Primary Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Cardiac MicroRNA Expression | before cardiopulmonary bypass and at 5 min after aortic de-clamping
  Samples were harvested from all the patients, respectively, before cardiopulmonary bypass and at 5 min after aortic de-clamping. Real-time quantitative stem-loop reverse transcription polymerase chain reaction assay was performed to detect the expression of microRNAs.

SECONDARY OUTCOMES:
Change from Baseline in Downstream Gene Expression | before cardiopulmonary bypass and at 5 min after aortic de-clamping
  Expressions of messenger RNAs and proteins were quantified for genes which are regulated by above-detected microRNAs.

CONTACTS AND LOCATIONS:
Overall Officials: Wanjun Luo, MD, Principal Investigator — Xiangya Hospital of Central South University
Locations (1):
- Xiangya Hospital, Changsha, Hunan, China

REFERENCES:
- [Derived] Gao Y, Huang R, Chen R, Li J, Luo W. Ischemic postconditioning altered microRNAs in human valve replacement. J Surg Res. 2016 Jan;200(1):28-35. doi: 10.1016/j.jss.2015.07.010. Epub 2015 Jul 10. PMID 26253453